CLINICAL TRIAL: NCT02683967
Title: The Impact of Acupuncture on the Success Rate of IVF Treatments
Brief Title: The Impact of Acupuncture on the Success Rates of IVF (In Vitro Fertilisation) Treatments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Homerton University Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: FE1303
Record Dates: First submitted 2016-01-11; First posted 2016-02-17 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture (Active Comparator): These patients received acupuncture during the follicular development phase and on the day of egg collection.
  Interventions: Procedure: acupuncture
- Control (No Intervention): Patients received standard care, no acupuncture.

INTERVENTIONS:
Procedure: acupuncture — patients received a Delphi acupuncture at least 3 times during their fertility treatment cycle.
  Arms: Acupuncture

SUMMARY:
The trial aims to investigate whether acupuncture has an effect in increasing clinical pregnancy (pregnancy that is confirmed by a scan) and live birth rates on women undergoing IVF treatment.

DETAILED DESCRIPTION:
Failing to conceive naturally poses significant stress to the infertile couple. It creates a feeling of failure and frustration. It has been found that the use of complementary therapies makes women feel empowered, with a sense of regaining control of the body.

The popularity of acupuncture is increasing. A significant proportion of couples having fertility treatment, especially IVF (In-Vitro Fertilisation) ask their clinician about using acupuncture and some patients undergo acupuncture privately without reporting to their clinicians.

The effectiveness of acupuncture on IVF has been extensively researched; however the results are varied and not conclusive. This is due to previous studies varying significantly in their study design, acupuncture timing and the final outcome measure. As a result of the difference in the studies it is not clear whether acupuncture is beneficial regarding IVF success rates and whether it should be offered to women undergoing IVF.

ELIGIBILITY:
Inclusion Criteria:

* Women under the age of 43 years with a BMI of less than 30 undergoing 1st or no more than their 2nd failed fresh IVF or ICSI cycle.

Exclusion Criteria:

* Those women undergoing frozen embryo replacement cycle or receiving donor eggs, BMI > 30 or currently having acupuncture/ any other form of CAM, having contraindication to acupuncture like those with HIV, Hep C will be excluded.

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 184 (Actual)
Dates: Start 2013-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Live birth rate | 18 months
  The primary objective is to determine the clinical effectiveness of acupuncture in improving live birth rates in women undergoing IVF

SECONDARY OUTCOMES:
Clinical pregnancy rate | 18 months
  The secondary objective is to determine whether acupuncture improves clinical pregnancy rate
Multiple pregnancy | 9 months
  To determine whether there is an increased rate of multiple pregnancy
Quality of life | 9 months
  To examine the effect of acupuncture on improving the quality of life for women by means of EQ% quality of life questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Karin Gillerman, Principal Investigator — NHS Honorary Contract

IPD SHARING:
Plan to Share IPD: No